CLINICAL TRIAL: NCT00478543
Title: Effect of Loop Diuretics Treatment on Blood Pressure Control in Phase 3-4 of Chronic Kidney Disease
Brief Title: Loop Diuretics in Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Giuseppe Conte, Chair of Nephrology Second University of Naples
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LD1-22052007
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Kidney Disease
Keywords: Loop diuretics; Chronic Kidney Disease; Hypertension; Blood pressure control; Left ventricular mass
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diuretic (Experimental): Furosemide
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide

SUMMARY:
The purpose of this study is to verify the efficacy of diuretic therapy on blood pressure control and left ventricular mass in patients affected by chronic kidney disease

DETAILED DESCRIPTION:
In CKD, impairment of renal function causes fluid and sodium retention and consequently expansion of extracellular volume, which corresponds to about 5% of body weight in absence of peripheral edema. In particular, sodium retention increases exponentially as glomerular filtration rate declines and is of primary importance in the pathogenesis of hypertension. Therefore, reduction of salt intake in renal patients allows a better blood pressure control. Despite the evidence collected on the beneficial effects of salt restriction in CKD, compliance with dietary prescription is generally poor in patients followed up in the real world of clinical practice. In the presence of poor adherence to salt restriction, diuretics agents become the cornerstone of treatment of hypertension secondary to CKD. Disappointingly, nephrologists are reluctant to "adequately" use loop diuretics in their hypertensive CKD patients, probably because of the fear of side effects and of the amazing absence in medical literature of studies of middle-long term on diuretic efficacy. Therefore, the primary aim of this study is to evaluate efficacy and safety of loop diuretics on blood pressure control in patients affected by CKD.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal insufficiency in stage CKD 3 and 4 (GFR 60-15 ml/min/m2) estimated by Cockcroft-Gault formula corrected for body surface
* Systolic blood pressure >140 mmHg in treatment with at least 1 class of antihypertensive drugs
* Patients not in treatment from at least one month with loop diuretics

Exclusion Criteria:

* Loop diuretics treatment
* Variation of serum creatinine >30% in the last 3 months
* Steroid therapy and/or cytotoxic agents
* Edema syndromes (Nephrotic syndrome, cirrhosis, heart failure NYHA class 3 or 4)
* Neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Attainment of blood pressure target (<130/80 mmHg)and evaluation of left ventricular mass by echocardiography | 6 months and 1 year respectively

SECONDARY OUTCOMES:
Adverse drug reactions, ambulatory blood pressure measure control, body volumes evaluated by bioimpedance analysis, expense of time and resources in follow-up of patients | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Conte, Professor, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- Nephrology Department, Second University of Naples, Naples, Italy

REFERENCES:
- [Background] De Nicola L, Minutolo R, Bellizzi V, Zoccali C, Cianciaruso B, Andreucci VE, Fuiano G, Conte G; investigators of the TArget Blood Pressure LEvels in Chronic Kidney Disease (TABLE in CKD) Study Group. Achievement of target blood pressure levels in chronic kidney disease: a salty question? Am J Kidney Dis. 2004 May;43(5):782-95. doi: 10.1053/j.ajkd.2004.01.009. PMID 15112168
- [Background] De Nicola L, Minutolo R, Chiodini P, Zoccali C, Castellino P, Donadio C, Strippoli M, Casino F, Giannattasio M, Petrarulo F, Virgilio M, Laraia E, Di Iorio BR, Savica V, Conte G; TArget Blood Pressure LEvels in Chronic Kidney Disease (TABLE in CKD) Study Group. Global approach to cardiovascular risk in chronic kidney disease: reality and opportunities for intervention. Kidney Int. 2006 Feb;69(3):538-45. doi: 10.1038/sj.ki.5000085. PMID 16395261
- [Background] Bellizzi V, Di Iorio BR, De Nicola L, Minutolo R, Zamboli P, Trucillo P, Catapano F, Cristofano C, Scalfi L, Conte G; ERIKA Study-group. Very low protein diet supplemented with ketoanalogs improves blood pressure control in chronic kidney disease. Kidney Int. 2007 Feb;71(3):245-51. doi: 10.1038/sj.ki.5001955. Epub 2006 Oct 11. PMID 17035939